CLINICAL TRIAL: NCT03989947
Title: A Phase 2 Open-Label Long-Term Extension Study to Evaluate the Safety and Efficacy of BMN 111 in Children With Achondroplasia
Brief Title: An Extension Study to Evaluate Safety and Efficacy of BMN 111 in Children With Achondroplasia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111-208
Record Dates: First submitted 2019-05-22; First posted 2019-06-18 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Achondroplasia
Keywords: Dwarfism; Bone Disease; ACH; Natriuretic Peptide C-Type; Musculoskeletal Diseases; Skeletal Dysplasias
MeSH Terms: conditions — Achondroplasia; Dwarfism; Bone Diseases; Musculoskeletal Diseases | interventions — vosoritide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active BMN 111 (Experimental): Once daily subcutaneous injections of recommended dose of BMN 111 based on weight-band dosing.
  Interventions: Drug: Active BMN 111: Subcutaneous injection of recommended dose of BMN 111 based on weight-band dosing once daily.

INTERVENTIONS:
Drug: Active BMN 111: Subcutaneous injection of recommended dose of BMN 111 based on weight-band dosing once daily. — Modified recombinant human C-type natriuretic peptide (subject to adjustment per protocol)
  Other Names: Vosoritide

SUMMARY:
This is a Phase 2, open-label multi-center long-term extension study, with approximately 70 subjects, to evaluate the safety and efficacy of BMN111 in children with Achondroplasia until subjects reach near-adult final height. Eligible subjects will have completed 1 year of BMN111 or placebo treatment in the 111-206 study and once enrolled in the 111-208 extension study will receive a daily dose of BMN111 by subcutaneous injection according to their age as determined by 111-206.

ELIGIBILITY:
Inclusion Criteria:

1. Must have completed Study 111-206 on investigational treatment (BMN 111 or placebo).
2. Parent(s) or guardian(s) are willing and able to provide written, signed informed consent after the nature of the study has been explained and prior to performance of any research related procedure. Also, subjects under the age of majority are willing and able to provide written assent (if required by local regulations or the IRB/IEC) after the nature of the study has been explained and prior to performance of any research-related procedure. Subjects who reach the age of majority in their country while the study is ongoing will be asked to provide their own written consent again upon reaching the legal age of majority.
3. Are willing and able to perform all study procedures

Exclusion Criteria:

1. Permanently discontinued BMN 111 or placebo prior to completion of Study 111-206
2. Have a clinically significant finding or arrhythmia on ECG that indicates abnormal cardiac function or conduction or QTc-F > 450 msec
3. Require any investigational agent (except BMN 111) prior to completion of study period
4. Current therapy with antihypertensive medications, angiotensin-converting enzyme (ACE) inhibitors, angiotensin II receptor blockers, diuretics, beta-blockers, calcium-channel blockers, cardiac glycosides, systemic anticholinergic agents, GnRH agonists, any medication that may impair or enhance compensatory tachycardia, diuretics, or other drugs known to alter renal or tubular function
5. Pregnant or planning to become pregnant (self or partner) at any time during the study
6. Concurrent disease or condition that, in the view of the investigator, would interfere with study participation or safety evaluations, for any reason
7. Have a condition or circumstance that, in the view of the investigator, places the subject at high risk for poor treatment compliance

Min Age: 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2038-05 (Estimated); Study Completion 2038-05 (Estimated)

PRIMARY OUTCOMES:
Evaluate the incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | "Through study completion, an average of 5 years"
  Number of study participants with treatment-emergent adverse events or serious adverse events
Evaluate change in height/length z-score in children with ACH treated with BMN 111 | "Through study completion, an average of 5 years"

SECONDARY OUTCOMES:
Evaluate the change from baseline of mean annualized growth velocity (AGV) | "Through study completion, an average of 5 years"
Characterize maximum concentration (Cmax) of BMN 111 in plasma | "Through study completion, an average of 5 years"
Characterize the area under the plasma concentration time-curve from time 0 to infinity (AUC0-∞) | "Through study completion, an average of 5 years"
Characterize the elimination half-life of BMN 111 (t½) | "Through study completion, an average of 5 years"
Characterize the apparent clearance of drug | "Through study completion, an average of 5 years"
Characterize the apparent volume of distribution based upon the terminal phase (Vz/F) | "Through study completion, an average of 5 years"
Characterize the amount of time BMN 111 is present at maximum concentration (Tmax) | "Through study completion, an average of 5 years"
Evaluate the change from baseline on body proportion ratios of the extremities | "Through study completion, an average of 5 years"
Effect of BMN 111 on bone morphology and quality by XRay | "Through study completion, an average of 5 years"
The effect of BMN 111 on bone morphology/quality will be assessed by measuring bone mineral density via Dual X-ray Absorptiometry | "Through study completion, an average of 5 years"
Potential Changes in health-related quality of life as measured by the quality of life in Short- statured youth | "Through study completion, an average of 5 years"
  Evaluate the long-term effect of BMN 111 on health-related quality of life, developmental status and functional independence, using age-specific QoL and functional independence questionnaires (Bayley-III, WeeFIM, ITQOL, QoLISSY, PedsQL, Child Behavior Checklist 1.5-5 [CBCL 1.5-5], Child Behavior Checklist 6-18 [CBCL 6-18]).
BMN 111 activity will be assessed by measuring bone and collagen metabolism | "Through study completion, an average of 5 years"
Describe the incidence of surgical and medical interventions related to achondroplasia | "Through study completion, an average of 5 years"
Assess effect on sleep disordered breathing by polysomnography in patients up to 5 years old. | "Through study completion, an average of 1 year"
Evaluate the effect of BMN 111 on skull and brain morphology, including foramen magnum, ventricular and brain parenchymal dimensions by MRI in patients up to 3 years old. | "Through study completion, an average of 1 year"

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director MD, Study Director — BioMarin Pharmaceutical
Locations (16):
- United States (9):
  - Children's Hospital & Research Center Oakland, Oakland, California
  - Harbor - UCLA Medical Center, Torrance, California
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Emory University, Decatur, Georgia
  - Ann Robert and H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Cincinnati Childrens Hospital, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Medical College of Wisconsin, Children's Hospital, Milwaukee, Wisconsin
- Australia (2):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Murdoch Children's Research Institute, Parkville, Victoria
- Japan (3):
  - Osaka University, Osaka
  - Saitama Children's Medical Center, Saitama
  - Tokushima University Hospital, Tokushima
- United Kingdom (2):
  - Guy's and St. Thomas NHS Foundation Trust Evelina Children's Hospital, London
  - Sheffield Children's NHS Foundation Trust, Sheffield